CLINICAL TRIAL: NCT03106792
Title: A Randomized, Double-blind, Placebo-controlled, 4-arm Parallel Study to Evaluate the Effectiveness of Hairfinity on Improving Hair Health and Rate of Growth
Brief Title: A Clinical Trial to Evaluate the Effectiveness of Hairfinity on Improving Hair Health and Rate of Growth
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brock Beauty Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 16HHHB
Record Dates: First submitted 2017-04-04; First posted 2017-04-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Hairfinity #1 (Experimental): Dosage form: Capsule Frequency: Take 2 capsules by mouth in the morning with a meal. Duration: 90 days
  Interventions: Dietary Supplement: Hairfinity #1
- Hairfinity #2 (Experimental): Dosage form: Capsule Frequency: Take 2 capsules by mouth in the morning with a meal. Duration: 90 days
  Interventions: Dietary Supplement: Hairfinity #2
- Hairfinity #3 (Experimental): Dosage form: Capsule Frequency: Take 2 capsules by mouth in the morning with a meal. Duration: 90 days
  Interventions: Dietary Supplement: Hairfinity #3
- Placebo (Placebo Comparator): Dosage form: Capsule Frequency: Take 2 capsules by mouth in the morning with a meal. Duration: 90 days
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Hairfinity #1 — Main Hairfinity formulation
  Arms: Hairfinity #1
Dietary Supplement: Hairfinity #2 — Variation to main formulation
  Arms: Hairfinity #2
Dietary Supplement: Hairfinity #3 — Variation to main formulation
  Arms: Hairfinity #3
Dietary Supplement: Placebo — No active ingredients
  Arms: Placebo

SUMMARY:
The primary outcome of the study is the effect of Hairfinity vs. Placebo on the rate of distal hair growth, assessed using Trichoscan HD, in healthy female adults from baseline to day 90 (end of study).

ELIGIBILITY:
Inclusion Criteria:

1. Female 18-50 years of age (inclusive)
2. Subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).

   OR

   Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include:
   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Intrauterine devices
   * Vasectomy of partner
   * Double Barrier Method
   * Non-heterosexual lifestyle
3. Fitzpatrick skin type of I-V (See appendix 3)
4. Willing to maintain the colour of and style of the hair cut for the duration of the study
5. Willing to maintain shampooing frequency and general hair regime for the duration of the study
6. Willing to not cut hair for the duration of the study
7. Willing to have area of hair prepped for Trichoscan analysis
8. Healthy as determined by laboratory results, medical history, and physical exam
9. Subjects must agree to comply with study procedures
10. Has given voluntary, written, informed consent to participate in the study

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant during the course of the trial.
2. Women who have begun hormonal birth control or hormone replacement within 6 months of randomization
3. Subjects taking natural health products, including multi-vitamins, botanicals and other nutraceuticals, within 2 weeks of randomization and for the duration of the study
4. Subjects with Fitzpatrick scores over V, which stems from the sensitivity of the testing method (requires a degree of color contrast when evaluating hair relative to skin)
5. Subjects having underwent a form of treatment for thinning hair, including prescription drugs or light therapy within 6 months of randomization
6. Medical history of diagnosed alopecia and/or trichotillomania (compulsive hair pulling). Medical history may be assessed by the Qualified Investigator
7. Subjects currently using hair extensions
8. Subjects with psoriasis or any active dermatological condition of the scalp at randomization that in the opinion of the qualified investigator would interfere with the clinical evaluations
9. Medical history of thyroid disorders or with TSH levels outside the normal range (0.4-4.5 ±0.05) as assessed by the Qualified Investigator
10. Unstable medical condition as determined by qualified investigator
11. Clinically significant abnormal lab results at screening will be assessed by the Qualified Investigator
12. History, or current diagnosis of any cancer (except for successfully treated basal cell carcinoma in an area other than the scalp) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission more than 5 years of diagnosis are acceptable.
13. Alcohol abuse or drug abuse within the past 6 months
14. Consumption of greater than 2 standard alcoholic drinks per day
15. Use of medicinal marijuana
16. Participation in a clinical research trial within 30 days prior to randomization
17. Allergy or sensitivity to study product and/or it's ingredients
18. Individuals who are cognitively impaired and/or who are unable to give informed consent
19. Any other condition which in the Investigator's opinion may adversely affect the subject's ability to complete the study or its measures or which may pose significant risk to the subject (e.g. cardiovascular, renal, lung, diabetes, psychiatric illness, bleeding disorders etc)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-06-29 (Actual); Study Completion 2018-06-29 (Actual)

PRIMARY OUTCOMES:
Rate of distal hair growth | 90 days
  assessed using Trichoscan HD

SECONDARY OUTCOMES:
Change in number of shed hair strands | 90 days
  assessed using the standardized wash test
Change in mean diameter of hair fibers | 90 days
  assessed using Trichoscan HD
Change in hair density | 90 days
  assessed using Trichoscan HD
Change in the number of terminal and vellus hairs | 90 days
  assessed using Trichoscan HD
Changes in the percent of hairs in the anagen and telogen phases | 90 days
  assessed using Trichoscan HD
Changes in hair quality parameters | 90 days
  assessed by a dermatologist
Changes in hair quality | 90 days
  assessed by a dermatologist
Changes in hair quality | 90 days
  assessed with self-assessment questionnaires

OTHER OUTCOMES:
Incidence of clinically significant abnormal vital signs | 90 days
Incidence of clinically significant abnormal complete blood panel | 90 days
Incidence of clinically significant abnormal electrolytes | 90 days
Incidence of clinically significant abnormal kidney function panel | 90 days
Incidence of clinically significant abnormal liver function panel | 90 days
Incidence of adverse events | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada